CLINICAL TRIAL: NCT05312944
Title: Polymyalgia Rheumatica Associated to Primary Sjogren Syndrome : A French Multicentric Retrospective Study (PASS)
Brief Title: Polymyalgia Rheumatica Associated to Primary Sjogren Syndrome
Acronym: PASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PASS (29BRC20.0176)
Record Dates: First submitted 2022-02-17; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Polymyalgia Rheumatica; Sjogren's Syndrome
MeSH Terms: conditions — Polymyalgia Rheumatica; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the phenotype of patients having PMR symptoms and primary Sjogren syndrome (pSS), we used a French national call to identify patients combining both diseases and collected retrospective clinical and biological data.

DETAILED DESCRIPTION:
A national call to identify patients combining pSS and PMR was disseminated in France. Patients with Sjögren's syndrome associated with rheumatoid arthritis were excluded. We described the global population having both diseases and compared them to two historic prospective cohorts of isolated pSS (the prospective cohort of primary Sjögren DiapSS), or isolated PMR (TENOR, a cohort of recent PMR), regarding clinical, imaging and treatments characteristics.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the ACR/EULAR 2012 criteria for PMR and the ACR/EULAR 2016 criteria for pSS

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients fulfilling the ACR/EULAR 2012 criteria for PMR and the ACR/EULAR 2016 criteria for pSS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
clinical data | at diagnosis
  pain (pain scale)
biological data | at diagnosis
  biology (CRP in mg/L)
biological data | at diagnosis
  presence of anti-SSA/SSB (yes/no)
histological data | at diagnosis
  accesories salivary glands biopsies (focus score)
imaging data | at diagnosis
  US (presence of shoulder involvement yes/no; hip involvement yes/no)
treatments data | at inclusion ( day 0)
  use of methotrexate yes/no; abatacept yes/no, rituximab yes/no, corticosteroids yes/no; pilocarpine yes/no; hydroxychloroquine yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France